CLINICAL TRIAL: NCT05027750
Title: Application Of The Theory Of Planned Behavior For Weight Control In Women: A Randomized Controlled Study
Brief Title: Theory-Based Obesity Intervention Program for Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, SEDA GOGER, Lecturer, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 162146620500104273
Record Dates: First submitted 2021-08-11; First posted 2021-08-30 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: obesity; women; health behaviors; Theory of Planned Behavior
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The selected womens were associated with obesity risk factors about obesity (overweight) or obese and between 18-49 years old) and randomly assigned to the experimental group. Obesity training consisting of a total of five sessions structured according to Theory of Planned Behavior was scheduled for the intervention group. Each session lasted for approximately 30 minutes.
  Interventions: Behavioral: Application of The Theory of Planned Behaviour For Weight Control
- Control (No Intervention): The control group of the Randomized Controlled Trial (RCT) was composed of 39 womens (between 18-49 years old) randomly assigned to the control group who are BMI was between 25.0-29.9 or BMI was between ≥30.0 according to the risk rating scales. A standard obesity training consisting of a single session was scheduled for the control group.

INTERVENTIONS:
Behavioral: Application of The Theory of Planned Behaviour For Weight Control — The training to be imparted to the participants was applied online in groups of 5-6 people via the Google Meet program. Obesity training consisting of a total of five sessions. Each session lasted for approximately 30 minutes. After the training given to intervention group, the women will be followed-up for 6 months. The women in the intervention group will be given counseling service by the researchers, and their status will be evaluated every month.
  Arms: Intervention

SUMMARY:
The aim of this study is to examine the effect of education and counseling given to women according to the Theory of Planned Behavior on weight management. This study will be conducted as a single-blind randomized controlled study consisting of intervention and control groups. A total of 78 overweight and obese women included in the study. The participants assigned to either of the groups by the block randomization method. A training program consisting of a total of five sessions applied to the intervention group, and counseling will be provided for 6 months. The data will be analyzed with Statistical Package for Social Sciences (SPSS) 22.0 package program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being a woman in the age group of 18-49 years
* Having a body mass index (BMI) of 25.0-30.0 kg/m2 (overweight) or >30.0 kg/m2 (obese)
* Not going through menopause
* Not having diabetes
* Not having thyroid disease
* Not using hormonal contraceptive pills
* Not having polycystic ovarian disease
* Not having a metabolic disease
* Not having Cushing's syndrome
* Not having a disease that prevents physical activity
* Not having hypertension
* Not being pregnant or breastfeeding
* Owning and using a smart phone
* Having a mail account in Google and being able to use it

Exclusion Criteria:

* Women who do not meet the inclusion criteria
* Not volunteering to participate in the study
* Women with communication problems
* Women who did not give consent at any stage of the study and who quit the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Healthy Lifestyle Behaviors-II Scale | 6 months
  Healthy Lifestyle Behaviors-II Scale aims to measure the health promotion behaviors of individuals. The scale consists of 52 items. It is a four-point Likert-type scale (1: "never," 2: "sometimes," 3: "often," and 4: "regularly"). The lowest score that can be obtained is 52, and the highest score is 208. High scores indicate that the individual practices the specified health behaviors at a high level.
International Physical Activity Questionnaire Short Form | 6 months
  International Physical Activity Questionnaire Short Form, the intensity (mild, moderate, and severe) of physical activity is taken into account to accommodate different types of physical activities. The questionnaire provides information about sitting, walking, and the time spent in moderately intense and vigorous activities. Vigorous physical activities have a value of 8.0 MET, moderate activities have a value of 4.0 MET, and walking has a value of 3.3 MET. The minute and frequency (day) values of the relevant activities are multiplied by the MET values. The total physical activity value is obtained by summing the multiplication values obtained at the last stage. Accordingly, the physical activity levels of individuals are classified as physically inactive (<600 MET-min/week), low physical activity (600-3000 MET-min/week), and adequate physical activity (health benefits) (>3000 MET-min/week).

SECONDARY OUTCOMES:
Change in body mass index | 6 months
  Weight and height will be combined to report BMI in kg/m^2. The change in body mass index will be evaluated.
Change in waist/hip ratio | 6 months
  Waist and hip will be combined to report Waist/Hip in cm. The change in waist/hip ratio will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Provincial Directorate of Health, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No